CLINICAL TRIAL: NCT06063642
Title: Real-time Functional Magnetic Resonance Imaging Neurofeedback Treatment for Young Adults With Internet Gaming Addiction
Brief Title: Neurofeedback for Internet Gaming Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Macau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSERE23-APP004-ICI
Record Dates: First submitted 2023-05-31; First posted 2023-10-02 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2023-09

CONDITIONS: Internet Gaming Disorder
Keywords: neurofeedback; behavior addiction
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Intervention Model Description: Eligible candidates will be randomly assigned to either receive the experimental feedback intervention or sham feedback intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants will be blind to the intervention group assignment until they complete the entire study procedure. An outcome assessor who is blind to this assignment will collect the primary outcome measurement data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental neurofeedback intervention (Experimental): In an approximately 30-minute training session, participants receive activity feedback from a midbrain region involved in reward processing and gaming addiction. Feedback will be presented in the form of a thermometer/bar in the middle of the screen and updated every two seconds. They will be trained to down-regulate the activity in this region with the help of this feedback using cognitive strategies. This down-regulation training is believed to be beneficial to addictive behaviors by the investigators.
  Interventions: Device: Neurofeedback training
- Sham feedback intervention (Sham Comparator): In an approximately 30-minute training session, participants receive activity feedback from a brain region irrelevant to reward processing or gaming addictive behavior. The feedback presentation form and task instructions will be the same as for the experimental group. Based on the functional role of the feedback region, the investigators do not believe this feedback training will change the addictive behaviors of the participants who receive this intervention.
  Interventions: Device: Sham feedback training

INTERVENTIONS:
Device: Neurofeedback training — Neurofeedback training is a type of non-invasive brain modulation technique that enables individuals to self-regulate brain activity patterns by providing them feedback on specific activity measures. Effective self-regulation is often linked to changes in cognition, behavior, and clinical symptoms.
  Arms: Experimental neurofeedback intervention
Device: Sham feedback training — A controlled form of neurofeedback training that provides feedback irrelevant to the targeted mental process.
  Arms: Sham feedback intervention

SUMMARY:
The primary aim of this study is to evaluate the therapeutic potential of real-time functional magnetic resonance imaging (MRI) neurofeedback in alleviating internet gaming disorder (IGD) symptoms by training individuals with such symptoms to down-regulate the activity in their reward-processing-related midbrain regions.

ELIGIBILITY:
Inclusion Criteria:

* Meet at least five of the Diagnostic and Statistical Manual of Mental Disorders fifth edition (DSM-5) criteria for IGD and score 38 or above on the Internet Addiction Test (IAT)
* First language is Chinese (Mandarin)
* Right-handed
* Have played the mobile game "King of Glory" for more than 3 years
* Ability to give informed consent
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Any primary diagnosis of a current psychological or neurological disorder
* Any history of psychological or neurological disorder
* Any MRI contraindication
* Currently on a psychotropic medication
* Any history of substance dependence
* Any history of brain injury or surgery

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in self-reported urge for internet gaming as assessed by Visual Analog Scales (1 to 100) | Up to 30 days after the intervention session

SECONDARY OUTCOMES:
Change in reward-related activity during exposure to internet gaming videos | Up to 3 days
  Participants will complete cue-reactivity tasks in which they are exposed to video clips captured from the dependent mobile game before and after the intervention. Functional MRI data will be collected to measure their pre- to post-intervention changes in the brain reward processing pathways.
Change in inhibitory response in the affective Go/Nogo task | Up to 3 days
  This task that uses affective Chinese characters as stimuli will be used to examine changes in inhibitory control performance as well as changes in brain activity associated with this cognitive process pre- to post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Yuan, Ph.D, Study Director — University of Macau
Locations (1):
- Centre for Cognitive and Brain Sciences, University of Macau, Taipa, Macau

REFERENCES:
- [Derived] Gu A, Chan CL, Xu X, Dexter JP, Becker B, Zhao Z. Real-Time fMRI Neurofeedback Modulation of Dopaminergic Midbrain Activity in Young Adults With Elevated Internet Gaming Disorder Risk: Randomized Controlled Trial. J Med Internet Res. 2025 Jan 29;27:e64687. doi: 10.2196/64687. PMID 39879613